CLINICAL TRIAL: NCT07350733
Title: Cognitive Training for First-Year Student Sleep and Wellness
Brief Title: Cognitive Training for Student Sleep and Wellness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, David Creswell, Co-Investigator, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP00012477
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Well-Being (Psychological Flourishing)
Keywords: Mindfulness; University Student; Sleep; Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Active Comparator): 14-day smartphone based mindfulness meditation training intervention consisting of a personalized introduction, a 10 to 15-minute audio-guided lesson, plus daily life homework practice (3-10 minutes) each day.
  Interventions: Behavioral: Equa
- Stress Management Training (Active Comparator): 14-day smartphone based training intervention focused on coping strategies consisting of a 10 to 15-minute audio-guided lesson, plus daily life homework practice (3-10 minutes) each day.
  Interventions: Behavioral: Coping Control

INTERVENTIONS:
Behavioral: Equa — Mindfulness for attention monitoring and acceptance with a focus on concentration, clarity, and equanimity
  Arms: Mindfulness Meditation
Behavioral: Coping Control — Problem-solving for cognitive coping
  Arms: Stress Management Training

SUMMARY:
This randomized control trial (RCT) explores two potential stress reduction interventions: a digital mindfulness program personalized for first year college students and a problem-solving based stress management program. These interventions were chosen because they rely on evidence-based approaches to stress management: problem-solving for cognitive coping and mindfulness for attention monitoring and acceptance with a focus on concentration, clarity, and equanimity. This selection allows for the assessment of the comparative efficacy of these methods in addressing student stress and stress-related outcomes (sleep duration, mental health, and academic success). Personalization to the college student offers the potential for greater engagement and user satisfaction by tailoring the program while maintaining the empirically driven structure of a digital mindfulness program. The investigators predict greater engagement and satisfaction will lead to higher adherence, and thus more skill-building. In this small RCT, first year college students will complete one of the two intervention conditions: Equa and MyTime. This will allow for the exploration of the effects of personalized mindfulness training compared to an active control condition.

This work has the potential for identifying effective, low-cost tools to help young adults manage their stress and stress-related health and may inform theory and future work on stress modification strategies for other populations. The main trials aims are:

Specific Aim 1. To explore whether a personalized mindfulness intervention (Equa) leads to greater adherence, engagement and use satisfaction compared to a digital stress management program.

Specific Aim 2. To explore whether a personalized mindfulness intervention leads to greater improvements in student stress and stress-related outcomes compared to a problem solving-based digital stress management program. Outcomes include perceived stress, depressive symptoms, nightly sleep duration, and grades.

DETAILED DESCRIPTION:
A sample of 100 first-year undergraduate students enrolled at Carnegie Mellon University will be recruited to participate in this study for the duration of the spring semester of 2026. Participants will be randomly assigned to complete 14-days of smartphone audio-guided lessons of either mindfulness (N=50) or a stress management program (N=50). Participants will complete baseline measures of stress, psychological well-being, and health behaviors. Participants will also be given a wearable device (FitBit) that will measures sleep and physical activity throughout the semester. For the 7 days prior to the intervention start and 7 days following the completed 14 day intervention, students will complete daily diaries that assess their thoughts, feelings, and experiences throughout the day. Participants will complete two more online surveys with similar questionnaires as the baseline assessment, one within 10 days of completing the intervention, and one at the end of the semester.

ELIGIBILITY:
Inclusion Criteria:

* Carnegie Mellon University undergraduate student in their 1st year of study
* 18 years of age or older
* Have a data-enabled smartphone
* Speak English
* On CMU's Pittsburgh campus for the duration of the Spring 2026 semester

Exclusion Criteria:

* Under 18 years of age at time of enrollment
* Not enrolled full-time as a student

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Adherence | From intervention program start at week 4 to end of treatment at week 6
  Number of lessons completed during the intervention period
App Engagement | From intervention program start at week 4 to end of treatment at week 6
  Self-reported measure of engagement following each lesson on a scale from 1-Not at all, to 5- Extremely.
User Satisfaction | From intervention program start at week 4 to end of treatment at week 6
  Self-reported user satisfaction with the intervention lesson measured on a scale of 1- Not at all, to 5- Extremely
Change in Self-Reported Perceived Stress | Change from baseline to post and 2-month follow-up
  The 10-item Perceived Stress Scale is a self-reported assessment of perceptions of stress over the past month. Total scores range from 0 to 40, with higher scores indicating higher levels of perceived stress.
Change in Self-Reported Depressive Symptomatology | Change from baseline to post and 2-month follow-up
  The Patient Health Questionnaire is an eight-item instrument that will be utilized as a brief measure of depression severity. A total score ranges from 0 to 24 and is calculated by adding each of the nine items' scores. A higher total score signifies more severe depression levels.
Total Nightly Sleep Duration | From study week 1 through 2-month follow-up
  Nightly sleep duration as measured in minutes by FitBit wearable devices.
Grade Point Average | From study week 1 through 2-month follow-up
  Student university cumulative grade point average calculated at the end of the semester.

SECONDARY OUTCOMES:
Change in Self-Reported Loneliness | Change from baseline to post and 2-month follow-up
  The UCLA Loneliness scale will be used to measure subjective feelings of loneliness and social isolation. A total score that ranges from 20 to 80 is calculated by summing the score of each item. A higher total score signifies increased feelings of loneliness.
Change in Self-Reported 2-way Social Support | Change from baseline to post and 2-month follow-up
  The 2-way social support scale will be used to assess experiences giving or receiving emotional and instrumental support. Total scores ranging from 0-60 and subscales (giving/receiving instrumental/emotional support) ranging from 0-15 are calculated , with a higher score indicating greater social support.
Change in Self-Reported Brief Resilience | Change from baseline to post and 2-month follow-up
  The brief resilience scale measures an individual's ability to bounce back from stress, adversity, and challenging life circumstances. An average is calculated across 6 items, with higher scores signifying greater brief resiliency. Scores can range from 1 to 5.
Change in Self-Reported Physical Health Symptoms | Change from baseline to post and 2-month follow-up
  The Cohen-Hoberman Inventory of Physical Symptoms assess how much 33 common physical symptoms have bothered or distressed an individual over the past two weeks from 0 (not bothered) to 4 (extremely bothered). Items are summed to create a composite score ranging from 0-132, with higher scores indicating more distress from physical symptoms.
Change in Self-Reported Sleep Quality | Change from baseline to post and 2-month follow-up
  The Pittsburgh Sleep Quality Index assess sleep quality over the past month. A global sleep quality score is calculated (ranging 0-21), with higher scores indicating worse sleep quality.
Change in Self-Reported Sleep Reactivity | Change from baseline to post and 2-month follow-up
  The Ford Insomnia Response to Stress Test is a 9-item measure of sleep reactivity. Participants rate how likely (1 - not likely, to 4 very likely) it is for them to have difficulty sleep in different scenarios, with total scores ranging from 9-36. Higher scores indicate greater stress-induced sleep reactivity.
Change in Self-Reported Anxiety | Change from baseline to post and 2-month follow-up
  The Generalized Anxiety Disorder 2-item scale measures anxiety symptoms over the past two weeks. Participants rate how bothered they have been by problems on a scale from 0 - not at all, to 3 - nearly every day. Scores are totaled to create a composite score, with higher scores indicating greater generalized anxiety.
Change in Engagement of Enjoyable Activities | Change from baseline to post and 2-month follow-up
  The Pittsburgh Enjoyable Activities Test is a brief, ten-item measure that will be used to assess the frequency of a participant's engagement in various activities on a scale of 0 (never) to 4 (every day). A total score ranges from 0 to 40 where a higher score reflects the increased frequency of participation in enjoyable activities.
Change in Self-Reported Mindfulness | Change from baseline to post and 2-month follow-up
  Evaluated using the The Five Facet Mindfulness Questionnaire, a 24-item scale measuring mindfulness. Each item is rated on a scale from 1=never or very rarely true to 5= very often or always true, with a higher total score indicating greater mindfulness tendencies.
Change in Self-Reported Social and Academic Fit | Change from baseline to post and 2-month follow-up
  The Sense of Social and Academic Fit Scale contains 17-items assessing perceptions of both social and academic fit. Participants respond from 1- Strongly Disagree to 7 - Strongly Agree, summed to create a composite score with higher values indicating higher feelings of belongingness.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided